CLINICAL TRIAL: NCT00614029
Title: A Randomized, Open-Label, Single-Dose, Four-way Crossover Study to Evaluate the Pharmacokinetics and Bioequivalence of Sumatriptan Delivered Via the Intraject System Versus IMITREX STATdose at Three Injection Sites in Healthy Adults
Brief Title: A Study to Evaluate the Pharmacokinetics and Bioequivalence of Sumatriptan Delivered Via the Intraject System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zogenix, Inc. (Industry)
Responsible Party: Stephen J. Farr, Ph.D/ President and COO, Zogenix, Inc
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ZX001-0601
Record Dates: First submitted 2008-01-07; First posted 2008-02-13 (Estimated); Last update posted 2022-11-10 (Actual); Status verified 2009-11

CONDITIONS: Pharmacokinetics; Bioequivalence
Keywords: sumatriptan; Injections; Subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A (Experimental): IMITREX -abd. to Intraject-abd. to IMITREX -thigh to Intraject-thigh
  Interventions: Device: Sumatriptan (via Intraject System)
- B (Experimental): Intraject-abd. to IMITREX -abd. to Intraject-thigh to IMITREX -thigh
  Interventions: Device: Sumatriptan (via Intraject System)
- C (Experimental): Intraject-abd to IMITREX -abd to Intraject-arm. to IMITREX -arm.
  Interventions: Device: Sumatriptan (via Intraject System)
- D (Experimental): IMITREX-abd to Intraject-abd to IMITREX-arm. to Intraject-arm.
  Interventions: Device: Sumatriptan (via Intraject System)
- E (Experimental): IMITREX-arm to Intraject-arm to IMITREX-thigh to Intraject-thigh
  Interventions: Device: Sumatriptan (via Intraject System)
- F (Experimental): Intraject-thigh to IMITREX-thigh to Intraject-arm to IMITREX-arm
  Interventions: Device: Sumatriptan (via Intraject System)

INTERVENTIONS:
Device: Sumatriptan (via Intraject System) — 0.5 mL of solution with 6 mg of sumatriptan (base) as the succinate salt

SUMMARY:
A study to evaluate the pharmacokinetics and bioequivalence of sumatriptan delivered by the Intraject system.

DETAILED DESCRIPTION:
A single center, randomized, single-dose, open-label, partial-block, four-period, four-way crossover study in 54 healthy adult subjects to evaluate the pharmacokinetics and bioequivalence of sumatriptan delivered by the Intraject system compared to IMITREX STATdose at three injection sites (abdomen, thigh, and arm.)

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Negative serum pregnancy test
* Female subjects of child-bearing potential must agree to use acceptable birth control 3 weeks prior to and 2 weeks after study dosing.
* Body Mass Index (BMI) and sufficient subcutaneous thickness, in the opinion of the investigator, for an injection into the abdomen, arm and thigh
* Non-tobacco user
* Adequate venous access in the left or right arm to allow collection of a number of blood samples
* Fluent in the English language
* Provide written informed consent to participate in the study and be willing to comply with the study procedures

Exclusion Criteria:

* History within the previous 2 years of drug or alcohol dependence
* Evidence of clinically relevant oral, cardiovascular, hematologic, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurologic, psychiatric or skin disorder
* History of epilepsy or other neurologic disease
* History of coronary disease, peripheral vascular disease, cerebrovascular accident, transient ischemic attack, uncontrolled hypertension, or signs/symptoms of ischemic heart disease
* History of allergy, anaphylaxis, or hypersensitivity to sumatriptan or similar drugs including sulphonamides
* History of scleroderma or any skin condition that may adversely affect the injection or absorption of subcutaneously administered medications
* Tattoos or birthmarks in the lateral thigh, abdominal area or arm (deltoid) that are large enough to restrict injection site selection and/or evaluation
* Positive screening test for HIV antibodies, Hepatitis B surface antigen, or Hepatitis C antibody
* Positive results on illicit drug test at Screening or at Check-in
* Use of any prescription medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2006-12; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-time curve, maximal plasma concentration, time to maximal concentration, terminal elimination half-life, and apparent terminal elimination rate constant of sumatriptan will be determined at each of 3 sites | one week

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Chandler, MD, Principal Investigator — Covance
Locations (1):
- Covance, Inc, Dallas, Texas, United States